CLINICAL TRIAL: NCT03132948
Title: Physical Activity and Quality of Life in Pediatric Patients With Acute Lymphoblastic Leukemia Receiving Maintenance Chemotherapy
Brief Title: Quality of Life in Pediatric Patients With Acute Lymphoblastic Leukemia Receiving Maintenance Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Principal Investigator, Andrea Orsey, Hematologist/Oncologist, Connecticut Children's Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-086
Record Dates: First submitted 2017-01-31; First posted 2017-04-28 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Quality of Life
Keywords: ALL Cancer Patients; Quality of Life; Fitness
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Physical Activity (Experimental): Single arm study where patients choose from physical activities after baseline assessment by PT. Activities include the following: Nintendo WII fit console, Xbox Kinect fit console and other sport activities.
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — Nintendo WII fit console, Xbox console, sport activities (soccer, basketball, yoga, walking and other physical games)

SUMMARY:
The purpose of the study is to evaluate the impact of exercise on physical activity levels and quality of life in children with acute lymphoblastic leukemia (ALL) receiving maintenance chemotherapy.

DETAILED DESCRIPTION:
Health-related quality of life is an important outcome of cancer treatment which encompasses physical, psychological, social, and functional well-being. In addition, quality of life includes one's overall ability to become a productive member of society and achieve personal fulfillment. Treatment of pediatric cancer is a highly stressful experience which can be challenging and disruptive to the lives of children and their families. Pediatric oncology patients receiving chemotherapy often experience a decline in quality of life due to decreased activity, fatigue, and psychological distress such as depression or anxiety when compared to healthy individuals. Preliminary data suggests that there is an association between physical activity and quality of life. Exercise has been show to improve mood, increase energy levels, and reduce stress. Although more research and clinical resources have been given to the effects of exercise on quality of life among adult cancer patients, there is a lack of research in these areas among children with cancer. The investigators know little about whether children with cancer would benefit from exercise.

The investigators have added a blood sample for biomarkers. Research in adult cancer patients have shown an association between different biomarkers and sleep quality which suggests that regulation of certain biomarkers may be affected through exercise in adults. Measures of biomarkers may provide insight into potential mediators between PA, sleep quality, or fatigue levels.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric oncology patients with ALL in the maintenance phase of chemotherapy during the time of study
* Ages 8-18 years of either gender (age limits due to reliability and validity of outcome assessment surveys)
* Have no documented or observable psychiatric or neurological disorders that would interfere with study participation
* Capable of speaking and reading English
* Having no contraindications to participate in moderate physical exercise as determined by the research staff and the patient's pediatric oncologist
* Currently living with their parents/legal guardians
* Consent obtained from legal guardians and assent obtained from patients to participate in the study

Exclusion Criteria:

* Not a pediatric oncology patient with ALL in maintenance
* Not receiving chemotherapy during the time of study
* Age less than 8 years or greater than 18 years
* Not English-speaking Since not all outcome measures have been validated in Spanish and other languages, only English-speaking patients will be included.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2010-10; Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Outcomes | 1 year
  PedsQL

SECONDARY OUTCOMES:
Physical Activity | 1 year
  Actigraphy
Sleep | 1 year
  Diary
Fatigue | 1 year
  Childhood Fatigue Scale

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Orsey, MD, Principal Investigator — Connecticut Children's Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
data will be de-identified to protect PHI
Supporting Information: Study Protocol, SAP, ICF
Time Frame: following completion of study for 5 years
Access Criteria: Researchers may contact PI